CLINICAL TRIAL: NCT01891734
Title: Enhancing Delivery of Problem Solving Therapy Using SmartPhone Technology
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PPO 13-122
Record Dates: First submitted 2013-06-25; First posted 2013-07-03 (Estimated); Results first posted 2016-09-16 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Depression; Anxiety
Keywords: Veterans; Health Services; Mental Health; Technology; Primary Health Care; Psychotherapy
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Problem Solving Therapy plus Moving Forward (PST-MF) (Experimental): All Veterans will receive a standard 6-session administration of Problem Solving Therapy (Nezu & D'Zurilla, 1999). Session 1 will take place in-person during a scheduled appointment and will last for 1 hour. Subsequent sessions will take place over the telephone and will last for approximately 30 minutes. Participants in this arm will also receive the Moving Forward app for SmartPhones, which was adapted from Problem Solving Therapy to be used either as a standalone treatment or as an adjunct to other related therapies such as in-person Problem Solving Therapy or the Moving Forward website. The phone content matches Problem Solving Therapy. Benefits of the app include 24-hours accessibility of psychoeducational materials and worksheets.
  Interventions: Other: Problem Solving Therapy plus Moving Forward
- Problem Solving Therapy (Active Comparator): All Veterans will receive a standard 6-session administration of Problem Solving Therapy (Nezu & D'Zurilla, 1999). Session 1 will take place in-person during a scheduled appointment and will last for 1 hour. Subsequent sessions will take place over the telephone and will last for approximately 30 minutes.
  Interventions: Other: Problem Solving Therapy

INTERVENTIONS:
Other: Problem Solving Therapy plus Moving Forward — All Veterans will receive a standard 6-session administration of Problem Solving Therapy (Nezu & D'Zurilla, 1999). Session 1 will take place in-person during a scheduled appointment and will last for 1 hour. Subsequent sessions will take place over the telephone and will last for approximately 30 minutes. Participants in this arm will also receive the Moving Forward app for SmartPhones, which was adapted from Problem Solving Therapy to be used either as a standalone treatment or as an adjunct to other related therapies such as in-person Problem Solving Therapy or the Moving Forward website. The phone content matches Problem Solving Therapy. Benefits of the app include 24-hours accessibility of psychoeducational materials and worksheets.
  Arms: Problem Solving Therapy plus Moving Forward (PST-MF)
Other: Problem Solving Therapy — All Veterans will receive a standard 6-session administration of Problem Solving Therapy (Nezu & D'Zurilla, 1999). Session 1 will take place in-person during a scheduled appointment and will last for 1 hour. Subsequent sessions will take place over the telephone and will last for approximately 30 minutes.
  Arms: Problem Solving Therapy

SUMMARY:
This project will be the first to evaluate the Moving Forward app in VA. Identifying an effective treatment for anxiety and depression in primary care is imperative within Veterans Health Administration as they are both common, chronic, and debilitating conditions associated with a number of personal and health-related costs. In close partnership with app developers at Mental Health Services, a major contribution of this research is the actionable feedback on the acceptability, feasibility and effectiveness of augmenting traditional Problem Solving Therapy with the Moving Forward app for future app development. If effectiveness can be established, Moving Forward has the potential for integration into the larger continuum of care for depression and anxiety in Primary Care-Mental Health Integration (e.g., care management, co-located collaborative care). Lastly, this pilot project will provide preliminary data for future research on SmartPhone technology. Veteran feedback on treatment components, ease of executing the study successfully and preliminary effect size calculations, will inform the design of the larger project.

DETAILED DESCRIPTION:
Access and engagement in evidence-based psychotherapies for Veterans are high priorities for the Veterans Health Administration, especially the Office of Rural Health and the office of Mental Health Services. SmartPhone applications are an emerging technology with a vast potential to extend the reach of traditional in-person psychotherapy by allowing increased digital access to providers and self-management tools. Due to the relatively recent development of this technology, there are no data on the effectiveness of SmartPhone-delivered psychotherapy. Preliminary data on acceptability and satisfaction are promising, suggesting a need for further research. The National Center for Posttraumatic Stress Disorder in collaboration with the National Center for Telehealth & Technology (T2) recently completed the development of an app called Moving Forward, a Veteran-friendly adaptation of Problem Solving Therapy, an evidence based therapy available through Primary Care Integration Clinics. In partnership with Mental Health Services, this proposed pilot project will gather preliminary data on the effectiveness and acceptability of Moving Forward and provide timely feedback to the app creators. Participants will include approximately 40 Veterans diagnosed with an anxiety or mood disorder interested in obtaining mental health treatment in Primary Care -Mental Health Integration. Participants will be randomly assigned to receive either Problem Solving Therapy augmented by the Moving Forward app or Problem Solving Therapy alone. Participants will complete assessments at baseline, 6 weeks and 12 weeks. Investigators propose 3 specific hypotheses. In hypothesis 1, investigators predict a moderate effect size will be observed when comparing homework completion and satisfaction for patients randomized to Problem Solving Therapy plus the Moving Forward app compared to patients randomized to Problem Solving Therapy alone. In hypothesis 2, investigators predict a moderate effect size will be observed when comparing change scores on the problem solving style for patients randomized to Problem Solving Therapy plus the Moving Forward app compared to patients randomized to Problem Solving Therapy alone. In hypothesis 3, investigators predict a moderate effect size will be observed when comparing depression, anxiety, stress and quality of life change for patients randomized to Problem Solving Therapy plus the Moving Forward app compared to patients randomized to Problem Solving Therapy alone. Key informant interviews will provide qualitative feedback on the Moving Forward app which investigators will share with our partners at Mental Health Services. The proposed project is important to the VA mission to improve access for all Veterans particularly those who face barriers to engagement in traditional face-to-face treatment. The proposed research addresses one of three primary focus areas of the Office of Research and Development (Access), two of Health Services Research &Development's research priorities (Access/Rural Health and Mental Health), and three of Secretary Shinseki's Transformational Initiatives for the 21st Century including improving: 1) access to care, 2) mental health, and 3) patient-centeredness. This proposed work is innovative as it focuses on a rapidly emerging mobile technology that has great potential to improve access and engagement in mental health service delivery. To date, there have been no randomized effectiveness trials that have examined SmartPhone apps for mental health service delivery. The project is also timely as there is a temporary moratorium (imposed by the Office of Information Technology) on app dissemination within Veterans Health Administration, presenting an opportunity to study Moving Forward prior to its release. At the completion of this project, investigators expect that the work proposed in this study will highlight the clinical value of the Moving Forward app, which will inform both VA policy makers and the scientific community at large about the utility of SmartPhone technology in mental health care delivery. Investigators also expect that this study will provide our partners at Mental Health Services with helpful feedback on the Moving Forward app design and future app development.

ELIGIBILITY:
Inclusion Criteria:

* Veterans will be eligible if they are 18 years old or older,
* speak and understand English,
* are patients in the Central Arkansas Veterans Healthcare System Primary Care-Mental Health Integration,
* and have a current diagnosis of depression

  * major depressive disorder, 296.2x and 296.3x
  * dysthymic disorder, 300.4
  * depressive disorder not otherwise specified, 311
* and/or anxiety

  * panic disorder without agoraphobia, 300.01
  * panic disorder with agoraphobia, 300.21
  * specific phobia, 300.29
  * social phobia, 300.23
  * obsessive-compulsive disorder; 300.3
  * posttraumatic stress disorder, 309.81
  * acute stress disorder, 308.3
  * generalized anxiety disorder, 300.02
  * anxiety disorder not otherwise specified, 300.00
* We considered enrolling only those Veterans diagnosed with mild-to-moderate depression, but chose to include a range of anxiety and depression-related disorders in order to reflect the population of Veterans seen in Primary Care-Mental Health Integration.
* Additionally, Problem Solving Therapy is designed to treat a range of stress-related problems, including both anxiety and depressive disorders.
* Veterans taking prescribed anxiolytics or anti-depressants will be eligible if they are on a stable medication regimen.

Exclusion Criteria:

* Exclusionary criteria include any current suicidal ideation,
* substance dependence diagnosis and current use,
* any psychotic spectrum diagnoses or
* inability to provide informed consent.
* Diagnosis will be confirmed by chart review and Mini International Neuropsychiatric Interview.
* Acute suicidal ideation will be determined by the assessing or treating clinician.
* During the baseline and follow-up interviews, any Veteran who endorses a "1" or higher on item # 21 on the Depression Anxiety and Stress Scale "I feel that life isn't worthwhile" or item # 9 on the Patient Health Questionnaire-9 "thoughts that you would be better off dead or of hurting yourself" will be asked follow-up questions on the suicide risk protocol (see appendix 3).
* Current substance or alcohol use will be determined by the alcohol and substance use modules of the Mini International Neuropsychiatric Interview.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Grubbs, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (1):
- Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Problem Solving Therapy-Moving Forward: Veterans in each group received 6-sessions of Problem Solving Therapy. Session 1 took place in-person immediately after the eligibility assessment and lasted for approximately 1 hour. Subsequent sessions took place over the telephone and lasted for approximately 30-45 minutes. As part of each PST session, participants completed the Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer & Williams, 2001) to evaluate on-going treatment effects and inquire about safety and suicidality. As part of the therapy, participants were asked to complete homework (psychoeducation about stress, information on effective problem solving and worksheets) using the Moving Forward app.
- Problem Solving Therapy: Veterans in each group received 6-sessions of Problem Solving Therapy. Session 1 took place in-person immediately after the eligibility assessment and lasted for approximately 1 hour. Subsequent sessions took place over the telephone and lasted for approximately 30-45 minutes. As part of each PST session, participants completed the Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer & Williams, 2001) to evaluate on-going treatment effects and inquire about safety and suicidality. As part of the therapy, participants were asked to complete homework (psychoeducation about stress, information on effective problem solving and worksheets) using the Moving Forward workbook.
Period: Overall Study
Arm/Group | Problem Solving Therapy-Moving Forward | Problem Solving Therapy
Started | 17 | 16
Completed | 14 | 13
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Population: Participants completed a demographic questionnaire, which inquired about age, race/ethnicity, gender, marital status, educational history, branch of military, war era, service connection, and familiarity with SmartPhone technology.
Groups:
- Total: Total of all reporting groups
Arm/Group | Problem Solving Therapy-Moving Forward | Problem Solving Therapy | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.12 (11.7) | 48.25 (12.7) | 46.64 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 14 | 12 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 7 | 10 | 17
  Black | 9 | 5 | 14
  Native American | 1 | 0 | 1
  Mixed Race | 0 | 1 | 1
Depression Anxiety and Stress Scale (DASS)-Depression [Mean (Standard Deviation); unit: units on a scale] — The 7-item depression subscale on the Depression Anxiety and Stress Scale (DASS) is measured on a 0-42 scale. Higher scores represent worse depression symptoms.
  units on a scale | 8.24 (4.87) | 9.25 (6.05) | 8.73 (5.41)
Depression Anxiety and Stress Scale (DASS)-Anxiety [Mean (Standard Deviation); unit: units on a scale] — The 7-item anxiety subscale on the Depression Anxiety and Stress Scale (DASS) is measured on a 0-42 scale. Higher scores represent worse anxiety symptoms.
  units on a scale | 6.65 (4.51) | 7.13 (5.83) | 6.88 (5.11)
Depression Anxiety and Stress Scale (DASS)-Stress [Mean (Standard Deviation); unit: units on a scale] — The 7-item stress subscale on the Depression Anxiety and Stress Scale (DASS) is measured on a 0-42 scale. Higher scores represent worse stress symptoms.
  units on a scale | 11.00 (4.03) | 11.19 (5.75) | 11.09 (4.86)
Short Form Health Survey-12-Veterans (SF-12 V) Mental Composite Score [Mean (Standard Deviation); unit: units on a scale] — The 12-item Short Form Health Survey-12-Veterans (SF-12 V) Mental Composite Score is rated on a 0-100 scale. Higher scores represent better mental health functioning.
  units on a scale | 36.98 (5.65) | 34.83 (6.07) | 35.94 (5.87)

OUTCOME MEASURES:

1. Primary Outcome: Depression Anxiety and Stress Scale (DASS)
Description: The 7-item depression subscale on the Depression Anxiety and Stress Scale (DASS) is measured on a 0-42 scale. Higher scores represent worse depression symptoms. The 7-item anxiety subscale on the Depression Anxiety and Stress Scale (DASS) is measured on a 0-42 scale. Higher scores represent worse anxiety symptoms. The 7-item stress subscale on the Depression Anxiety and Stress Scale (DASS) is measured on a 0-42 scale. Higher scores represent worse stress symptoms.
Time Frame: 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Problem Solving Therapy-Moving Forward | Problem Solving Therapy
Number analyzed (Participants) | 17 | 16
units on a scale
  DASS-Depression week 6 | 6.14 (5.76) | 5.23 (5.15)
  DASS-Anxiety week 6 | 7.21 (4.53) | 5.62 (4.59)
  DASS-Stress week 6 | 11.29 (6.59) | 8.23 (5.31)
  DASS-Depression week 12 | 6.14 (5.76) | 5.23 (5.15)
  DASS-Anxiety week 12 | 7.21 (4.53) | 5.62 (4.59)
  DASS-Stress week12 | 11.29 (6.59) | 8.23 (5.31)

2. Secondary Outcome: Short Form Health Survey-12-Veterans (SF-12 V) Mental Composite Score
Description: The 12-item Short Form Health Survey-12-Veterans (SF-12 V) Mental Composite Score is rated on a 0-100 scale. Higher scores represent better mental health functioning.
Time Frame: 6 weeks, 12 weeks
Population: These data include all participants who completed the 6-week follow-up assessment. Two participants from the PST-MF group did not complete the 6-week follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Problem Solving Therapy Plus Moving Forward (PST-MF): All Veterans will receive a standard 6-session administration of PST (Nezu & D'Zurilla, 1999). Session 1 will take place in-person during a scheduled appointment and will last for 1 hour. Subsequent sessions will take place over the telephone and will last for approximately 30 minutes. Participants in this arm will also receive the Moving Forward app for SmartPhones, which was adapted from PST to be used either as a standalone treatment or as an adjunct to other related therapies such as in-person PST or the Moving Forward website. The phone content matches PST. Benefits of the app include 24-hours accessibility of psychoeducational materials and worksheets.
  Problem Solving Therapy plus Moving Forward: All Veterans will receive a standard 6-session administration of PST (Nezu & D'Zurilla, 1999). Session 1 will take place in-person during a scheduled appointment and will last for 1 hour. Subsequent sessions will take place over the telephone and will last for approximately 30 minutes
- Problem Solving Therapy: All Veterans will receive a standard 6-session administration of PST (Nezu & D'Zurilla, 1999). Session 1 will take place in-person during a scheduled appointment and will last for 1 hour. Subsequent sessions will take place over the telephone and will last for approximately 30 minutes.
  Problem Solving Therapy: All Veterans will receive a standard 6-session administration of PST (Nezu & D'Zurilla, 1999). Session 1 will take place in-person during a scheduled appointment and will last for 1 hour. Subsequent sessions will take place over the telephone and will last for approximately 30 minutes.
Arm/Group | Problem Solving Therapy Plus Moving Forward (PST-MF) | Problem Solving Therapy
Number analyzed (Participants) | 15 | 16
units on a scale
  SF-12 V-Mental Composite Score 6 weeks | 40.00 (6.77) | 37.19 (7.50)
  SF-12 V Mental Composite Score 12 weeks | 39.92 (8.93) | 40.15 (10.89)
Statistical Analysis 1: Comparison: Problem Solving Therapy Plus Moving Forward (PST-MF) vs Problem Solving Therapy; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Cohen's d = .30

3. Secondary Outcome: Client Satisfaction Questionnaire (CSQ-8)
Description: The 8-item Client Satisfaction Questionnaire (CSQ-8) is rated on an 8-32 scale. Higher scores represent greater satisfaction with the intervention.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Problem Solving Therapy Plus Moving Forward (PST-MF) | Problem Solving Therapy
Number analyzed (Participants) | 17 | 16
units on a scale | 27.87 (3.36) | 29.06 (2.62)
Statistical Analysis 1: Comparison: Problem Solving Therapy Plus Moving Forward (PST-MF) vs Problem Solving Therapy; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Cohen's d = 0.30

ADVERSE EVENTS:
Time Frame: Participants were enrolled in the study for 12 weeks (3 months). Adverse events were monitored throughout their study participation.
Arm/Group | Problem Solving Therapy Plus Moving Forward (PST-MF) | Problem Solving Therapy
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No